CLINICAL TRIAL: NCT06240793
Title: Comparison of Unilateral and Bilateral Transforaminal Epidural Steroid Injection in Unilateral Lumbosacral Disc Herniation: a Randomized Controlled Trial
Brief Title: Comparison of Unilateral and Bilateral Transforaminal Epidural Steroid Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hanzade Aybuke Unal, Medical Doctor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/267
Record Dates: First submitted 2024-01-14; First posted 2024-02-05 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Pain, Chronic
Keywords: pain
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral transforaminal epidural block (Other): The necessary oblique and cranio-caudal angles will be provided in fluoroscopy for the patients' designated procedure area. Skin and subcutaneous tissue anesthesia will be applied to the injection site with 3 ml of 2% prilocaine. The neural foramen will be entered using a blunt-tipped sympathetic block needle and a guiding needle. After needle localization is confirmed with antero-posterior and lateral fluoroscopic images, 1-2 ml of contrast material will be injected following negative aspiration. After confirming the contrast material spread in the anterior epidural area and periradicular area, 8 mg dexamethasone will be injected. If the application will be performed bilaterally, the specified techniques will be applied in half the same way on the bilateral side. Patients will be observed for one hour after the procedure for possible complications.
  Interventions: Procedure: unilateral transforaminal epidural steroid block
- bilateral transforaminal epidural block (Active Comparator): The necessary oblique and cranio-caudal angles will be provided in fluoroscopy for the patients' designated procedure area. Skin and subcutaneous tissue anesthesia will be applied to the injection site with 3 ml of 2% prilocaine. The neural foramen will be entered using a blunt-tipped sympathetic block needle and a guiding needle. After needle localization is confirmed with antero-posterior and lateral fluoroscopic images, 1-2 ml of contrast material will be injected following negative aspiration. After confirming the contrast material spread in the anterior epidural area and periradicular area, 8 mg dexamethasone will be injected. If the application will be performed bilaterally, the specified techniques will be applied in half the same way on the bilateral side. Patients will be observed for one hour after the procedure for possible complications.
  Interventions: Procedure: bilateral transforaminal epidural steroid block

INTERVENTIONS:
Procedure: unilateral transforaminal epidural steroid block — unilateral transforaminal epidural steroid block
  Arms: Unilateral transforaminal epidural block
Procedure: bilateral transforaminal epidural steroid block — bilateral transforaminal epidural steroid block
  Arms: bilateral transforaminal epidural block

SUMMARY:
Lumbar radicular pain affects the person's quality of life. The most common cause of lumbar radicular pain is disc herniation. In radicular pain due to lumbar disc herniation, epidural steroid injections are frequently applied to patients who do not benefit from medical treatment and physical medicine modalities. Epidural steroid injection inhibits the synthesis and release of pro-inflammatory substances that develop as a result of mechanical compression.In the transforaminal epidural technique, the solution is administered to the anterior epidural space and spreads to the ipsilateral periradicular area. The applied solution does not cross the midline and there is no contralateral drug spread. Although bilateral transforaminal epidural steroid injection is recommended in unilateral lumbosacral disc herniation because the inflammation is bilateral, unilateral transforaminal steroid injection has been applied in most studies. We aimed to to evaluate the effects of unilateral and bilateral transforaminal epidural steroid injection on pain intensity, functionality and medication use in unilateral lumbosacral disc herniation

DETAILED DESCRIPTION:
Lumbar radicular pain is a condition that is very common The lifetime incidence of lumbar radicular pain is up to 43%. The most common cause of lumbar radicular pain is disc herniation. Other reasons; spinal stenosis, tumor, infection, spondylosis, spondylolisthesis, ligamentum flavum hypertrophy and synovial cyst. Lumbar disc herniation is most commonly located at L4-5 and L5-S1. Nerve compression due to disc herniation can occur in the spinal canal, lateral recess, neuroforaminal or extraforaminal region.

Inflammatory and mechanical reactions between the intervertebral disc, posterior longitudinal ligament and nerve roots play a role in the development of radicular pain. Chemical mediators released from the herniated disc increase the inflammatory response, and prostaglandin is released due to phospholipase A2 production. This situation results in radicular pain. Epidural steroid injections are frequently applied to patients in the treatment of radicular pain who do not benefit from medical treatment (non-steroidal anti-inflammatory analgesic, opioid, gabapentin, pregabalin) and physical medicine modalities. Epidural steroid injections can be administered via interlaminar, transforaminal or caudal routes. Epidural steroid injection inhibits the synthesis and release of pro-inflammatory substances that develop as a result of mechanical compression. In the transforaminal technique, the solution is administered to the anterior epidural space and spreads to the ipsilateral periradicular area. The applied solution does not cross the midline and there is no contralateral drug spread. In interlaminar epidural steroid injection, the solution crosses the midline and spreads bilaterally; but it remains in the posterior epidural area. Injection applied to the anterior epidural area adjacent to the nerve root via the transforaminal route is target-specific and a more effective form of treatment. In a study researchers reported that there was a greater decrease in pain intensity in patients with spinal stenosis with bilateral transforaminal epidural injection compared to interlaminar epidural injection. In another study, transforaminal injection was found to be superior in pain palliation compared to interlaminar injection in symptomatic lumbar disc herniation. Although there are studies in the literature comparing the advantages of epidural injection methods in lumbar disc herniation, there are no studies comparing the clinical effect of unilateral and bilateral transforaminal injection. Although bilateral transforaminal epidural steroid injection is recommended in unilateral lumbosacral disc herniation because the inflammation is bilateral, unilateral transforaminal steroid injection has been applied in most studies. (9- This study aims to evaluate the effects of unilateral and bilateral transforaminal epidural steroid injection on pain intensity, functionality and medication use in unilateral lumbosacral disc herniation and to observe whether they are superior to each other.

A single-center, prospective randomized controlled study will be conducted at Ankara University Faculty of Medicine, Department of Algology. Within the scope of the study, patients with radicular pain radiating to the unilateral lower extremities due to lumbosacral disc herniation will be evaluated with Magnetic Resonance Imaging (MRI) and physical examination between 1.6.2023 and 1.10.2023. The study included patients between the ages of 18 and 65, who had unilateral lumbosacral radicular pain for at least 3 months, whose MRI and physical examination confirmed lumbosacral disc herniation, who developed pain secondary to unilateral lumbosacral disc herniation, who did not respond to conservative treatment (medical and physical medicine modalities), and 128 patients with pain intensity of 4 and above measured using Numeric Rating Scala (NRS) will be included. Patients with previous lumbar surgery, patients with psychiatric illnesses who are unstable/not controlled by medical treatment, pregnant patients, patients with bleeding diathesis, patients who have received epidural steroid injection within the last year, patients who are exposed to substances given during the procedure (local anesthetic, steroid, contrast material). Patients with known allergies, scoliosis, spondylolisthesis, central canal stenosis, compression fracture, previous discitis, sequestered disc, and bilateral disc herniation will be excluded from the study.

Patients will receive epidural steroid injection through a unilateral or bilateral transforaminal approach. Within the scope of the study, patients with unilateral lumbosacral disc herniation and who are deemed suitable for transforaminal epidural steroid injection will be numbered in the order they are included in the study. Patients given an odd number will receive unilateral transforaminal epidural steroid injection, and patients given an even number will receive bilateral transforaminal epidural steroid injection. Transforaminal epidural steroid injections will be administered by Hanzade Aybüke Ünal. Pre-procedure and post-procedure evaluations of the patients will be recorded by Ahmet Basari, who is blind to the procedure performed. Demographic information of the patients, including age, gender, comorbidities, pain duration, and disc herniation level, will be recorded before the procedure. Before the procedure, pain intensity will be evaluated using the NRS 11 scale, and functionality will be evaluated using the ODI. The amount of medication used by the patients (non-steroidal anti-inflammatory analgesics, opioids, gabapentin, pregabalin) will also be noted. Patients will be contacted by phone at 1st week, 1st month and 3rd month to obtain information about NRS and ODI. During the specified time periods, pain intensity will be recorded using the NRS 11 scale, functionality will be recorded using the ODI, and medication use (non-steroidal anti-inflammatory analgesic, opioid, gabapentin, pregabalin) will be recorded. Additionally, possible complications in patients will also be recorded. A 50% or more reduction in pain intensity will be considered a response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65
* Patients with unilateral lumbosacral radicular pain for at least 3 months
* Lumbosacral radicular pain is confirmed by Magnetic Resonance Imaging (MRI) and physical examination and the pain is secondary to unilateral lumbosacral disc herniation.
* Patients who did not respond to conservative treatment (medical and physical medicine modalities)
* Pain intensity measured using Numeric Rating Scala (NRS) is 4 or more

Exclusion Criteria:

* Patients with previous lumbar surgery
* Presence of psychiatric disease that is unstable/not controlled by medical treatment
* Pregnant patients
* Those with bleeding diathesis
* Patients who received epidural steroid injection within the last year
* Patients with known allergies to the substances administered during the procedure (local anesthetic, steroid, contrast material)
* Patients with scoliosis, spondylolisthesis, central canal stenosis, compression fracture, previous discitis, sequestered disc, bilateral disc herniation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
pain severity | 3 months
  In patients who received unilateral and bilateral transforaminal steroid injection, pain severity change by using Numeric Ratin Scala was observed 3 months after the procedure.

SECONDARY OUTCOMES:
functionality | 3 months
  We evaluated the effect of unilateral and bilateral transforaminal epidural steroid injection on functionality in a 3-month period using the Oswestry Disability Index.
medication use | 3 months
  We evaluated the effect of unilateral and bilateral transforaminal epidural steroid injection on medication use in a 3-month period
Complication | 3 months
  We detected complications of unilateral and bilateral transforaminal epidural steroid injection application in a 3-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Hanzade A Unal, MD, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Germann C, Gotschi T, Sutter R. Predictive value of immediate pain relief after lumbar transforaminal epidural injection with local anesthetics and steroids for single level radiculopathy. Skeletal Radiol. 2022 Oct;51(10):1975-1985. doi: 10.1007/s00256-022-04051-3. Epub 2022 Apr 8. PMID 35394165
- [Background] Konstantinou K, Dunn KM. Sciatica: review of epidemiological studies and prevalence estimates. Spine (Phila Pa 1976). 2008 Oct 15;33(22):2464-72. doi: 10.1097/BRS.0b013e318183a4a2. PMID 18923325
- [Background] Lee JH, An JH, Lee SH. Comparison of the effectiveness of interlaminar and bilateral transforaminal epidural steroid injections in treatment of patients with lumbosacral disc herniation and spinal stenosis. Clin J Pain. 2009 Mar-Apr;25(3):206-10. doi: 10.1097/AJP.0b013e3181878f9e. PMID 19333170
- [Background] Liu J, Zhou H, Lu L, Li X, Jia J, Shi Z, Yao X, Wu Q, Feng S. The Effectiveness of Transforaminal Versus Caudal Routes for Epidural Steroid Injections in Managing Lumbosacral Radicular Pain: A Systematic Review and Meta-Analysis. Medicine (Baltimore). 2016 May;95(18):e3373. doi: 10.1097/MD.0000000000003373. PMID 27149443
- [Background] Makkar JK, Gourav KKP, Jain K, Singh PM, Dhatt SS, Sachdeva N, Bhadada S. Transforaminal Versus Lateral Parasagittal Versus Midline Interlaminar Lumbar Epidural Steroid Injection for Management of Unilateral Radicular Lumbar Pain: A Randomized Double-Blind Trial. Pain Physician. 2019 Nov;22(6):561-573. PMID 31775403
- [Background] Schaufele MK, Hatch L, Jones W. Interlaminar versus transforaminal epidural injections for the treatment of symptomatic lumbar intervertebral disc herniations. Pain Physician. 2006 Oct;9(4):361-6. PMID 17066121
- [Derived] Unal HA, Basari A, Ozgencil BK, Ozgencil GE, Erkoc SK. Comparison of Unilateral and Bilateral Transforaminal Epidural Steroid Injections in Unilateral Lumbar Disc Herniation: A Randomized Controlled Trial. J Clin Med. 2024 Dec 30;14(1):147. doi: 10.3390/jcm14010147. PMID 39797230